CLINICAL TRIAL: NCT06824961
Title: Does Increasing the Compression Pause From 3 to 5 Seconds in Mechanical Compression Devices Increase Ventilation Success Rate and Return of Spontaneous Circulation?
Acronym: LUCASVP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Prof. Dr. Patrick Schober, Principal Investigator: Professor Emergency Medicine in Anesthesiology Dr. Patrick Schober, MD, PhD., Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LUCASVP
Record Dates: First submitted 2025-01-21; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Arrest (CA)
Keywords: Advanced life support; Basic life support; Cardiac arrest; Cardiopulmonary resuscitation; CPR; ALS; BLS; Out-of-hospital cardiac arrest; OHCA; Mechanical chest compression devices; Mechanical CPR; Ventilation
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Multicenter, single blinded (patients), randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention - 5-second ventilation pause (Experimental): Patients in this group will have ventilation pauses lasting 5 seconds in between cardiac compressions given by mechanical CPR
  Interventions: Other: 5-second ventilation pause duration during mechanical CPR
- Control - 3-second ventilation pauses (Active Comparator): Patients in this group will have ventilation pauses lasting the standard 3 seconds in between cardiac compressions given by mechanical CPR
  Interventions: Other: 3-second ventilation pause duration during mechanical CPR

INTERVENTIONS:
Other: 5-second ventilation pause duration during mechanical CPR — The intervention is a 5-second lasting ventilation pause during mechanical CPR
  Arms: Intervention - 5-second ventilation pause
Other: 3-second ventilation pause duration during mechanical CPR — The intervention is a 3-second lasting ventilation pause during mechanical CPR
  Arms: Control - 3-second ventilation pauses

SUMMARY:
To give chest compressions during cardiopulmonary resuscitation (CPR), mechanical chest compression devices can be used. During synchronous 30:2 CPR, the standard setting on these devices leave an automated 3-second chest compression pause after 30 compressions to facilitate caregivers in providing two ventilations. With this standard setting, research has shown that in less than half of ventilation pauses during CPR, those two ventilations are given. Increasing the ventilation pause duration to 5 seconds instead of 3 seconds is also an option following current guideline recommendations, and aligns with measured ventilation pause duration in manual CPR. Increasing pause duration to 5 seconds could result in an increased ventilation success rate. This multicenter randomized controlled trial will randomize LUCAS® mechanical compression devices to a standard setting of 3- or 5-second compression pauses. The main outcome will be the percentage of ventilation pauses in which two ventilations are successfully given. Secondary outcomes include the restoration of spontaneous circulation (ROSC), and the difference in (neurologically intact) survival. No study has been performed to evaluate this effect yet.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥16 years of age)
* OHCA patients with an attempt at cardiopulmonary resuscitation (CPR) by ambulance personnel
* LUCAS® 3.1 has been used during the resuscitation attempt

Exclusion Criteria:

* Missing ambulance run report, missing or unclear impedance signal (measurement of resistance across the thorax), making it impossible to assess the number of ventilation pauses
* Absence of a minimum of 3 assessable pauses intended for ventilation after connecting the LUCAS®

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 692 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of ventilation pauses in which two ventilations are given | From enrollment to end of mechanically assisted CPR by ambulance nurses (approximate maximum timeframe of 3 hours)
  The difference in percentage of ventilation pauses in which two ventilations are given between the intervention and control group

SECONDARY OUTCOMES:
Return of spontaneous circulation (ROSC) | From enrollment to end of cardiac arrest treatment (approximate maximum timeframe of 5 hours)
  The difference in percentage of participants with and without ROSC
Cerebral performance score (CPC score) at hospital discharge (CPC 1-2 vs. 3-4) | From enrollment to hospital discharge (approximate maximum timeframe of 3 months)
  The difference in percentage of participants with a CPC of 1-2 (good neurological recovery) vs. 3-4 (poor neurological recovery) at hospital discharge
  CPC score system:
  1. Normal (good cerebral performance)
  2. Moderate disability (disabled but independent)
  3. Severe disability (conscious but disabled and dependent)
  4. Unconscious (coma or vegetative state)
Survival to hospital discharge | From enrollment to hospital discharge (approximate maximum timeframe of 3 months)
  The difference in percentage of participants with and without survival to hospital discharge
30-day survival | From enrollment to 30 days after cardiac arrest
  The difference in percentage of participants with and without survival at 30 days after the cardiac arrest
Number of rhythm checks per five minutes, expected | From enrollment to prehospital termination of CPR or handover at hospital by ambulance nurses (approximate maximum timeframe of 3 hours)
  The difference in the number of rhythm checks per five minutes performed with and without pausing the mechanical compression device, compared to the expected number of rhythm checks in that time frame (once every two minutes) between groups
Number of rhythm checks per five minutes, observed | From enrollment to prehospital termination of CPR or handover at hospital by ambulance nurses (approximate maximum of 3 hours)
  The difference in the number of rhythm checks per five minutes performed with and without pausing the mechanical compression device, compared to the observed number of rhythm checks in that time frame (once every two minutes) between groups
Average tidal volume (ml) | From enrollment to end of intra-arrest ambulance monitor registration or flow/pressure measurements (approximate maximum timeframe of 3 hours)
  Difference in average tidal volumes (ml) between groups
Average minute volume (ml/min) | From enrollment to end of intra-arrest ambulance monitor registration or flow/pressure measurements (approximate maximum timeframe of 3 hours)
  Difference in average minute volumes (ml/min) between groups
Average respiratory rate (rate per minute) | From enrollment to end of intra-arrest ambulance monitor registration or flow/pressure measurements (approximate maximum timeframe of 3 hours)
  Difference in average respiratory rate (rate per minute) between groups
Average airway pressure (cmH2O) | From enrollment to end of intra-arrest ambulance monitor registration or flow/pressure measurements (approximate maximum timeframe of 3 hours)
  Difference average airway pressures (cmH2O) between groups
Chest compression fraction (CCF) | From enrollment to end of intra-arrest registration of ambulance monitor (approximate maximum timeframe of 3 hours)
  Difference in chest compression fraction (CCF) between groups
Subjective experience of ambulance nurses with the mechanical CPR device and it's ventilation pause settings | After the last inclusion of the study, with an approximate time frame of 1-2 months to respond to the anonymous survey
  Exploratory anonymous questionnaire of subjective experience of ambulance nurses with the mechanical CPR device (the LUCAS) and it's ventilation pause settings during the resuscitation.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schober, MD, PhD, Principal Investigator — Amsterdam UMC
Locations (2):
- Netherlands (2):
  - Ambulance Amsterdam, Amsterdam, North Holland
  - Regionale Ambulance Voorziening Kennemerland - Ambulancezorg GGD Kennemerland, Haarlem, North Holland

IPD SHARING:
Plan to Share IPD: Undecided